CLINICAL TRIAL: NCT04067856
Title: Intravitreal Dexamethasone Implant (Ozurdex) Versus Bevacizumab in Patients With Diabetic Macular Edema Undergoing Cataract Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Allergan (Industry); Doheny Image Reading Center (Other)
Responsible Party: Principal Investigator, Pradeep Prasad, Assistant Clinical Professor of Ophthalmology, UCLA, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22361-01
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Macular Edema; Cataract
MeSH Terms: conditions — Cataract | interventions — Bevacizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevacizumab (Active Comparator): Intravitreal injection of 1.25mg/0.05cc bevacizumab
  Interventions: Drug: Bevacizumab Injection
- Dexamethasone implant (Active Comparator): Intravitreal injection of 0.7mg dexamethasone implant
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Bevacizumab Injection — Intravitreal injection
  Other Names: dexamethasone implant injection

SUMMARY:
The purpose of this research is to compare the effectiveness of bevacizumab (Avastin) with another a dexamethasone implant (Ozurdex), with respect to anatomic and visual outcomes as well as injection frequency in subjects undergoing cataract surgery with a concurrent diagnosis of diabetic macular edema (DME).

DETAILED DESCRIPTION:
Subjects over the age of 18 with both: 1) visually significant cataracts requiring cataract surgery and 2) diabetic macular edema (DME) will be enrolled in the study. Subjects with high risk proliferative diabetic retinopathy and any other retinal vascular disease or retinal pathology that may limit vision will be excluded. Baseline photography will be done to quantify the amount of DME and to exclude the presence of proliferative diabetic retinopathy or other retinal vascular or general retinal pathology. Subjects will be randomized to receive either an intravitreal injection of Ozurdex or Avastin at the time of cataract surgery. Subjects will be monitored the day after surgery, one to two weeks after cataract surgery and again monthly thereafter for a total of six visits from the time of cataract surgery with standardized visual acuity measurement, ophthalmologic examination and retinal photography performed at each visit. For the first two months after cataract surgery, subjects receiving Ozurdex will receive an injection of Avastin if the degree of swelling worsens by more than 10% on photography or the vision decreases. For the first two months after cataract surgery, subjects receiving Avastin will receive repeat injections of Avastin on a monthly basis. For each monthly visit thereafter, both groups will receive an intravitreal injection of Avastin if clinically significant DME is present or if vision declines.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old with type one or type two diabetes mellitus
* Center-involving diabetic macular edema with central subfield thickness ≥ 320um on Heidelberg Spectralis optical coherence tomography (OCT) testing
* Best-corrected electron-early treatment diabetic retinopathy study (E-ETDRS Visual Acuity) visual acuity letter score between 78 to 24
* Any Lens Opacities Classification System (LOCS) III cataract grade greater than or equal to two

Exclusion Criteria:

* Presence of macular edema attributable to other causes including but not limited to retinal venous occlusive disease and non-infectious uveitis
* History of glaucoma
* History of steroid-induced intraocular pressure (IOP) elevation that required IOP-lowering treatment
* Optic nerve cup to disc ratio greater than 0.6
* Active proliferative diabetic retinopathy
* Presence of other retinal diseases including but not limited to age-related macular degeneration, retinal venous occlusive disease and posterior segment uveitis
* Any prior intraocular surgery
* Treatment with any anti-VEGF medication within the past 3 months or intravitreal steroid within the past 6 months
* Panretinal photocoagulation within the prior 6 months or anticipated need for panretinal photocoagulation within the next 6 months
* IOP greater than or equal to 25
* Systolic blood pressure > 180 mmHg or diastolic > 110 mmHg
* Myocardial infarction, other cardiac event requiring hospitalization, cerebrovascular accident, transient ischemic attack or treatment for acute congestive heart failure within the past 6 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Final visual acuity | 6 month

SECONDARY OUTCOMES:
Final optical coherence tomography central macular thickness | 6 month
Total number of intravitreal injections over study period | 6 month

IPD SHARING:
Plan to Share IPD: No